CLINICAL TRIAL: NCT02895152
Title: The Role of Activity Monitors in Improving Physical Activity in COPD Patients Participating in Pulmonary Rehabilitation
Brief Title: Activity Monitor Use in COPD Patients Undergoing Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 197737
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic Bronchitis
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Activity Monitors; Fitbit; Fitness Tracker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Experimental): Those randomised to the feedback arm will receive weekly feedback on their activity levels and tailored advice on how to improve activity levels.
  Interventions: Behavioral: Feedback
- Control (No Intervention): Control arm will wear the activity monitor as specified in the protocol but will not receive feedback on activity levels

INTERVENTIONS:
Behavioral: Feedback — Will receive feedback on the amount of activity that has been undertaken in the last week, will specialist advice on steps taken, active minutes each day, how much device has been worn and tailored advice on how to improve activity levels
  Arms: Feedback

SUMMARY:
In patients with Chronic Obstructive Pulmonary Disease (COPD) lifestyles with lower physical activity levels have been shown to increase the risk of hospital admissions and shorten survival rates. An established process in increasing activity levels is to undergo pulmonary rehabilitation classes.

The investigators wish to identify whether the use of activity monitors,which will provide feedback on activity levels, will increase the physical activity levels of patients with COPD outside of the supervised pulmonary rehabilitation sessions.

DETAILED DESCRIPTION:
The research proposal has been developed in conjunction with the Respiratory Physicians and Physiotherapy team who deliver the pulmonary Rehabilitation sessions.

The investigators want to address if providing patients with monitors to record activity levels and then giving feedback on activity level data enhances the effect of the standard pulmonary rehabilitation program. The investigators want to pay particular attention to the levels of activity outside the duration of the rehabilitation classes - to see if higher levels of activity are reached.

This aims to be a feasibility study done on a small scale where issues such as compliance with wearing the device can be monitored closely. Compliance will be reviewed during a one week trial of wearing the device prior to starting the rehabilitation sessions. It will also enable study participants to get into the routine of wearing the device, charging etc.

Analysis of the data will be data collected during weekdays, choosing the 4 weekdays where there is a minimum of 8hrs of wearing time during waking hours. If the device has been worn for less than 8 hours, then days with most wear-time of the device will be selected. This method was chosen as it is a robust and statistically validated method of assessing activity levels in patients with COPD.

All study participants will be asked to wear the activity monitor to minimise any bias in the collected data. Subjects will be randomised as to whether they receive feedback or not.

The choice of activity monitor to be used was considered. Requirements are that it should be wrist-worn and the data collected by the device able to been downloaded through the associated computer software/"app". Wrist worn devices were chosen so that compliance in wearing the device would be maximized - they are worn in the same way a normal wrist watch would be.

A model from the brand "Fitbit" was selected based on this criteria. This was justified by previous studies showing Fitbit has good validity and usability in measuring energy expenditure in COPD patients.

As all participants in the study will partake in the pulmonary rehabilitation sessions there will be no deviations from standard care with this project. Analysis of activity will be downloaded, once a week, from the devices during the sessions and subjects randomised to receive feedback will have a 10 minute session dedicated to this.

There is a risk that subjects will have an exacerbation of their condition/chest infection during the period of pulmonary rehab. If a subject is too unwell to attend a rehabilitation session they will receive their feedback on their next attendance. Any subjects that are hospitalised during the study will be withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COPD diagnosis with spirometry: Forced expiratory volume at one second (FEV1)/Forced Vital Capacity (FVC) <70%
* Optimised pharmacology intervention
* Referred for Pulmonary Rehabilitation

Exclusion Criteria:

* FEV1 <30% predicted
* Clinical instability - Exacerbation in preceding 6 weeks
* Other clinical condition that prevents mechanical exercise (and therefore participation in sessions) due to pain/discomfort (Arthritis etc.)
* None compliant with the use of the activity monitors. Compliance will be assessed during the 1 week before starting the pulmonary rehabilitation programme (at the same time of collecting baseline data on activity). Compliance will be defined as wearing the activity monitors for at least 85% of the time allowing for times to take it off for charging.
* Recurrent chest infections >3 in the past 12 months.
* Unable to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Daily physical activity measured as: A: number of minutes active during the day; B: number of steps* | Through Study completion, upto 7 weeks total
  from the data recorded on the device

SECONDARY OUTCOMES:
Assessment of exercise capacity: 6 minute walk test (comparing the 2 groups and in comparison to baseline) | At beginning and at 7 weeks, with repeat at 6 months
Self reported exercise diary - duration of exercise | Through Study completion, upto 7 weeks total
Self reported exercise diary - BORG (perceived activity levels and effort scale) | Through Study completion, upto 7 weeks total
Assessment of symptom severity using Copd Assessment Test (comparing the 2 groups and in comparison to baseline) | Through Study completion, upto 7 weeks total
Assessment of symptom severity using Hospital Anxiety and Depression Scale (comparing the 2 groups and in comparison to baseline) | Through Study completion, upto 7 weeks total
Assessment of symptom severity using the Patient Activation Measure Score (comparing the 2 groups and in comparison to baseline) | Through Study completion, upto 7 weeks total
Assessment of symptom severity using the Chronic Respiratory Disease Questionaire Score (comparing the 2 groups and in comparison to baseline) | Through Study completion, upto 7 weeks total

CONTACTS AND LOCATIONS:
Overall Officials: Nawar D Bakerly, MD, FRCP, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Salford Royal NHS Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No